CLINICAL TRIAL: NCT07098910
Title: Surfactant Therapy Via Supraglottic Airway Device Versus Endotracheal Intubation to Prevent Mechanical Ventilation in Preterm Neonates With Respiratory Distress Syndrome: An Open-label, Non-inferiority, Randomized Controlled Trial at a Level-III Neonatal Intensive Care Unit in Vietnam
Brief Title: Surfactant Therapy Via Supraglottic Airway to Preterm Neonates With RDS in Vietnam
Acronym: NEOSURF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Göteborg University (Other); University of Padova (Other); Hanoi Obstetrics and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Tobias Alfvén, Professor of Global Child Health, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2089 CN/PS; Project-ID 2018-02770 VR (Other Grant/Funding Number: Swedish Research Council); RS2020-0 (Other Grant/Funding Number: ALF Region Stockholm); ALFGBG-998065 (Other Grant/Funding Number: ALF Region Västra Götaland); 2-4435/2024 (Other Grant/Funding Number: Carl Bennet AB)
Record Dates: First submitted 2025-07-21; First posted 2025-08-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: surfactant therapy; supraglottic airway device; laryngeal mask airway; preterm infant; neonate; newborn; vietnam; SALSA; RDS; respiratory distress syndrome; very low birth weight
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome | interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, single-centre, two-arm parallel-group, open-label, non-inferiority RCT with a 1:1 allocation ratio per neonate. The trial entails an internal pilot-phase of the first 100 patients.
Masking Description: The trial statistician conducting the final analysis will be masked to intervention arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surfactant therapy administered via supraglottic airway device (SALSA) (Experimental): Study participants will receive surfactant therapy via a preterm size supraglottic airway device (SALSA).
  Interventions: Procedure: Surfactant Administration Through Laryngeal or Supraglottic Airways (SALSA)
- Endotracheal intubation - surfactant administration - and extubation (INSURE) (Active Comparator): Study participants will receive surfactant therapy administered via brief endotracheal intubation - surfactant administration - and extubation (INSURE).
  Interventions: Procedure: Intubation - Surfactant administration - Extubation (INSURE)

INTERVENTIONS:
Procedure: Surfactant Administration Through Laryngeal or Supraglottic Airways (SALSA) — While the infant is spontaneously breathing on nasal CPAP, the NICU physician will place the supraglottic airway device (SAD) and assess airway adequacy via CO₂ detection, chest movement, bilateral breath sounds, gastric insufflation, oxygen saturation, and heart rate. Each placement attempt should last no more than 30 seconds, with up to two attempts allowed. Surfactant (Curosurf 200 mg/kg) will be given slowly in 1-2 ml aliquots via a CE-marked preterm-sized SAD, Neo i-gel® (sizes 0.85, 0.75, 0.65; Intersurgical Ltd). The infant should primarily breathe spontaneously with PEEP from a T-piece resuscitator and receive gentle PPV if needed. PPV is continued for 30 seconds after surfactant administration before SAD removal. A reservoir bag may be used secondarily to provide PPV. If surfactant delivery via SALSA fails, the INSURE method (Intubation-Surfactant-Extubation) will be attempted.
  Other Names: Laryngeal mask airway surfactant administration; Surfactant Therapy via Laryngeal Mask Airway; Laryngeal Mask Airway for Surfactant Administration in Neonates; Supraglottic airway devices for surfactant treatment
  Arms: Surfactant therapy administered via supraglottic airway device (SALSA)
Procedure: Intubation - Surfactant administration - Extubation (INSURE) — Study participants will receive surfactant therapy administered via brief endotracheal intubation - surfactant administration - and extubation (INSURE). Infants will be ventilated using a T-piece resuscitator with PEEP of 6 cm H20 and positive pressure ventilation (20 cm H20) for a couple of minutes (no more than 15 minutes) with adjustable FiO2. No mechanical ventilation will be used. Secondarily a reservoir-bag will be used for ventilation.
  Arms: Endotracheal intubation - surfactant administration - and extubation (INSURE)

SUMMARY:
Preterm babies often have trouble breathing because their lungs are not fully developed. This condition is called respiratory distress syndrome (RDS). A medicine called surfactant helps their lungs open up and work better. It is usually given through a procedure called INSURE, where a breathing tube is placed into the baby's trachea (via an endotracheal tube) to deliver the medicine. While effective, this method is invasive and can be uncomfortable and risky for the baby.

A newer, less invasive method called SALSA uses a soft mask placed in the throat (a laryngeal mask airway) instead of an endotracheal tube to give the surfactant. This randomized controlled trial will compare SALSA to the traditional INSURE method to see if it works just as well in preventing the need for invasive breathing support within three days of treatment.

The study will include preterm babies born before 34 weeks of pregnancy and weighing at least 750 grams, at Phu San Hanoi Hospital in Vietnam. If SALSA is found to be safe and effective, it may offer a gentler, less invasive, and easier-to-perform option for treating respiratory distress syndrome in premature babies.

DETAILED DESCRIPTION:
BACKGROUND

Respiratory distress syndrome (RDS) remains a leading cause of morbidity and mortality among preterm infants worldwide. Surfactant replacement therapy has significantly improved outcomes; however, standard techniques such as INSURE (Intubation-Surfactant-Extubation), while effective in avoiding mechanical ventilation, require endotracheal intubation-a procedure associated with potential complications and demanding considerable clinical expertise. Less invasive methods, such as surfactant administration via a laryngeal mask airway (SALSA), have shown promising results in reducing the need for mechanical ventilation in moderately preterm infants in smaller studies. This approach may be particularly beneficial in low- and middle-income countries (LMICs), where high birth volumes and limited availability of skilled personnel and advanced respiratory support highlight the need for simpler, safer interventions.

Evidence for SALSA in more immature preterm populations and from large randomized controlled trials remains limited. One key barrier to broader adoption has been the lack of appropriately sized supraglottic airway devices for very small infants. A recent feasibility study by this research team, using newly available preterm-sized devices, demonstrated that SALSA is feasible for surfactant delivery in infants weighing between 750 and 1500 grams (NCT06606444). A randomized controlled trial is now warranted to assess the effectiveness and safety of SALSA, particularly in lower-middle-income settings and among extremely low birth weight infants.

AIM AND HYPOTHESIS

This trial primarily aims to evaluate whether surfactant administration via the SALSA method is non-inferior to the current standard INSURE method in preventing IMV in preterm neonates with RDS admitted to a tertiary-level neonatal unit in South-Easia. It also seeks to compare the two methods in terms of safety, ease of use, infant comfort during the procedure, and morbidity during hospital admission.

We hypothesize that in preterm neonates with RDS, born before gestational week 34 and with a birth weight of at least 750 grams (P), surfactant administration via SALSA (I) will be non-inferior to INSURE (C) in preventing invasive mechanical ventilation (IMV) (O) within 72 hours after the procedure (T).

TRIAL DESIGN

This is an investigator-initiated, single-centre, two-arm parallel-group, open-label, non-inferiority RCT with a 1:1 allocation ratio per neonate. The trial entails an internal pilot-phase of the first 100 patients.

PARTICIPANTS:

See Eligibility section.

STUDY SITE

Phu San Hanoi Hospital (PSH) is the largest obstetric hospital in Hanoi, Vietnam, with about 40 000 deliveries every year and about 10% preterm births. The neonatal department is divided into three units: a level III NICU (35 beds), a high dependency unit (60 beds), and a Kangaroo mother care (KMC) unit (45 beds) which are staffed by 73 nurses and 21 doctors. Head ultrasound is made within 7 days of life and before discharge for all preterm infants <32 weeks of gestation as routine care, with additional assessments in between as needed. Echocardiography to screen for persistent ductus arteriosus is performed in neonates with clinical signs and treated medically (ibuprofen or paracetamol) if found haemodynamically significant. All infants <32 weeks of gestation are routinely examined for retinopathy of prematurity by ophthalmologist.

STUDY PROCEDURE

All infants requiring surfactant therapy will be screened for eligibility by the NICU team on a continuous basis. Caregivers will be approached for informed consent prior to inclusion. Eligible infants with consent will be randomized immediately before surfactant administration using a computer-generated, block-randomized sequence to receive either SALSA (intervention) or INSURE (control). The interventions are described in detail under "Arms and Interventions." For SALSA, a CE-marked, supraglottic airway device, Neo i-gel®, available in three sizes 0.85, 0.75, and 0.65 (Intersurgical Ltd), will be used. Procedural data will be collected through direct observation by the clinical team, while background characteristics and follow-up variables will be extracted from medical records by the study team. All data will be entered into an electronic case report form (eCRF) in REDCap. A subset of 50 patients per treatment arm will be video-recorded and reviewed for detailed analysis of procedure duration, physiologic stability and pain.

OUTCOMES

The primary outcome is: Failure of surfactant therapy to prevent invasive mechanical ventilation within 72 hours after first surfactant administration.

Decision to initiate mechanical ventilation via intubation will be made at the discretion of the treating physician, guided by the local NICU criteria for mechanical ventilation.

Secondary outcomes are listed under Outcome Measures.

SAMPLE SIZE

According to a baseline study conducted in 2023 (unpublished data), we assume that 21,5% of neonates in the control group (INSURE) would meet failure criteria. If there is no difference between SALSA and INSURE in terms of use of IMV (21,5% in both arms), 418 neonates need to be enrolled to be 80% sure that the upper limit of a one-sided 95% confidence interval will exclude an absolute difference larger than 10% in favour of INSURE. The sample is increased to 440 neonates to take into account a dropout of 5%.

PILOT PHASE

The trial will begin with an internal pilot phase designed to assess the feasibility of recruitment, adherence to trial procedures, data completeness, and intervention fidelity. Efficacy will not be evaluated. The internal pilot phase will enrol 100 neonates (approximately 23% of the total sample size), with recruitment anticipated over 12 months. This design will allow feedback on recruitment capacity and process quality and enabling adaptations.

The pilot phase will assess outcomes related to recruitment feasibility, adherence to intervention, adherence to mechanical ventilation criteria, retention, data completeness, data integrity and acceptability. Pilot outcomes are listed under Outcome Measures.

An interim assessment will be performed after the enrolment of 50 participants or after 12 months, whichever comes first. Only pilot outcomes will be assessed. The final analysis of the pilot phase will take place upon completion of enrolment of 100 participants. Following this evaluation, the Trial Steering Committee will determine whether to continue the study without modifications, implement protocol amendments-such as the inclusion of additional trial sites or adjustments to trial procedures-or temporarily suspend the trial to allow for a redesign. These decisions will be guided by a balanced assessment across all pilot domains.

ELIGIBILITY:
Inclusion Criteria:

* Inborn neonate (=born in the hospital), AND
* Gestational age <34+0 weeks, AND
* Birth weight ≥750g, AND
* Age <48 hours, AND
* Diagnosis of RDS, confirmed with a chest x-ray or lung ultrasound, except in cases where immediate treatment is necessary and imaging would cause a delay AND
* Indication for surfactant treatment: Infant on non-invasive support (CPAP/NIPPV) and FiO2 >0.30 to maintain oxygen saturation (SpO2) between 90% and 95%

Exclusion Criteria:

* Severe respiratory insufficiency in need of intubation at delivery room
* Severe respiratory insufficiency in need of intubation and invasive mechanical ventilation after arrival to NICU
* Previous surfactant administration
* Previous invasive mechanical ventilation
* Known pneumothorax
* Major malformations
* Physician not confident with study intervention
* The physician decided not to include the patient due to a preference for performing INSURE
* Excluded due to time constraints preventing completion of informed consent and trial procedures

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Failure of surfactant therapy to prevent invasive mechanical ventilation | Within 72 hours after first surfactant administration
  Categorical variable (Yes/No). Failure in terms of the need for endotracheal intubation and invasive mechanical ventilation. Decision to initiate mechanical ventilation via intubation will be made at the discretion of the treating physician, guided by the local NICU criteria for mechanical ventilation. Data is extracted from medical records.
  Analysis considerations:
  * If an infant deteriorates after randomization and requires intubation with mechanical ventilation before the allocated intervention can be performed, the case will be classified as failure in the intention-to-treat (ITT) analysis, but excluded from the per-protocol (PP) analysis.
  * If an infant improves after randomization and the allocated intervention is not required, the case will be included and not considered a failure in the ITT analysis, but excluded from the PP analysis.

SECONDARY OUTCOMES:
Early failure of surfactant therapy | Within 1 hour after first surfactant administration
  Categorical variable (Yes/No). Defined as use of invasive mechanical ventilation within 1 hour of first surfactant administration. Data is collected from medical record.
Late failure of surfactant therapy | Between 1 hour and 72 hours after first surfactant administration
  Categorical variable (Yes/No). Defined as use of invasive mechanical ventilation. Data is collected from medical record.
Time to initiation of invasive mechanical ventilation after the procedure | Before discharge (about 6-15 weeks)
  Numerical variable. Elapsed time between procedure initiation and mechanical ventilation, derived from medical record timestamps.
Invasive mechanical ventilation at any time during admission | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Decision to initiate mechanical ventilation via intubation will be made at the discretion of the treating physician, guided by the local NICU criteria for mechanical ventilation. Data is extracted from medical records.
Incidence of severe bradycardia | During the procedure, an average of 5-10 minutes
  Defined as <60 beats per minute. Measured by pulse oximetry and noted by team performing procedure.
Incidence of severe desaturation | During the procedure, an average of 5-10 minutes
  Defined as SpO2 <70%. Measured by pulse oximetry and noted by team performing procedure.
Change in FiO₂ (%) from before the procedure to 3 hours after surfactant administration | Within 10 minutes before the procedure to 3 hours after first surfactant administration
  Numerical variable. Observed by clinical team and noted in CRF.
Number of placement attempts needed to place LMA or ETT | During the procedure, an average of 5-10 minutes
  Numerical variable. Placement attempt defined as LMA or ETT entering the mouth with intent to place device in the airway. Observed by clinical team during procedure and noted in CRF.
Failure to place supraglottic airway device (SAD) or endotracheal tube (ETT) at first attempt | During the procedure, an average of 5-10 minutes
  Categorical variable (Yes/No). Failure to place device (SAD or ETT) and obtain an adequate airway on first attempt, as assessed by treating physician.
Volume of postintervention surfactant-resembling gastric residuals | Directly after first surfactant administration
  Numerical variable (ml). Gastric residuals are aspirated before procedure and directly after procedure (after SAD or ETT is removed) and volume of fluid content resembling surfactant is observed by clinical team and noted in CRF.
Proportion (%) of postintervention gastric surfactant aspirated of total surfactant dose | Directly after first surfactant administration
  Numerical variable (%). Fraction (calculated from residual aspirated surfactant and total dose (mL). Observed by clinical team during procedure and noted in CRF.
Postintervention gastric surfactant aspirated greater than 10% of surfactant dose | Directly after first surfactant administration
  Categorical variable (Yes/No). Calculated from ratio below 10% from Proportion (%) of postintervention gastric surfactant aspirated. Observed by clinical team during procedure and noted in CRF.
Reflux of surfactant during procedure | Directly after first surfactant administration
  Categorical variable (Yes/No). Clinical reflux of surfactant during procedure. Observed by clinical team during procedure and noted in CRF.
Number of surfactant doses given during admission | Before discharge (about 6-15 weeks)
  Numerical variable. Number of surfactant doses. Data is collected from medical record.
Administration of a second surfactant dose within 6 hours of the first dose | 6 hours after initial dose
  Categorical variable (Yes/No). Data is collected from medical record.
Method of subsequent surfactant doses | Before discharge (about 6-15 weeks)
  Method used for delivery of subsequent surfactant doses. Data is collected from medical record.
Incidence of mortality within 7 days after birth | Seven days of age
  Categorical variable (Yes/No). Data is collected from medical record.
Incidence of mortality prior to discharge | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Data is collected from medical record.
Time to death | Before discharge (about 6-15 weeks)
  Numerical variable. Elapsed time between birth and death. Derived from medical record notations.
Duration of invasive mechanical ventilation | Before discharge (about 6-15 weeks)
  Numerical variable (days). Data is collected from medical record.
Duration of Continuous Positive Airway Pressure (CPAP) or Non-invasive Positive Pressure Ventilation (NIPPV) | Before discharge (about 6-15 weeks)
  Numerical variable (days). Data is collected from medical record.
Duration of any respiratory support (IMV, CPAP, NIPPV or oxygen by nasal cannula) | Before discharge (about 6-15 weeks)
  Numerical variable (days). Data is collected from medical record.
Duration of hospital admission | Before discharge (about 6-15 weeks)
  Numerical variable (days). Data is collected from medical record.
Incidence of bronchopulmonary dysplasia | 36 weeks post menstrual age
  Categorical variable (Yes/No). Defined as need for oxygen or ventilatory support for at least 28 days and persisting at 36 weeks of postmenstrual age (ventilatory support: IMV, CPAP/NIPPV or O2 by nasal cannula). Data is collected from medical record.
Postnatal steroid treatment before discharge | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Data is collected from medical record.
Incidence of IVH grade III or IV | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Head ultrasound is made within 7 days of life and before discharge for all preterm infants <32 weeks of gestation (and older infants with complications) as routine care, with additional assessments in between as needed. Data is collected from medical record.
Incidence of cystic periventricular leukomalacia | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Head ultrasound is made within 7 days of life and before discharge for all preterm infants <32 weeks of gestation (and older infants with complications) as routine care, with additional assessments in between as needed. Data is collected from medical record.
Incidence of pneumothorax, requiring drainage | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Pneumothorax requiring drainage by needle thoracocentesis or chest drain. Data is collected from medical record.
Incidence of pulmonary haemorrhage, requiring circulatory support | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Defined as pulmonary haemorrhage requiring circulatory support like fluid bolus, blood transfusion or vasopressors/inotropes. Data collected from medical records.
Incidence of persistent ductus arteriosus requiring treatment | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Requiring medical (ibuprofen or paracetamol) or surgical treatment. Data is collected from medical record.
Incidence of early-onset sepsis | Within 72 hours after birth.
  Defined by clinical signs, laboratory findings, or positive blood culture, as assessed by the treating clinician within 72 hours of birth. Data is collected from medical record.
Incidence of late-onset sepsis | >72 hours after birth to discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Defined by clinical signs, laboratory findings, or positive blood culture, as assessed by the treating clinician from 72 hours after birth to discharge. Data is collected from medical record.
Incidence of retinopathy of prematurity, ≥ grade 3 | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). All infants <32 weeks of gestation are assessed by Ophthalmologists as clinical routine. Data is collected from medical record.
Incidence of transfer due to need of intestinal surgery | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Eg. need of surgery due to necrotizing enterocolitis, spontaneous intestinal perforation or ileus. All cases with indication for surgery are referred to the neighbouring Vietnam National Children's Hospital. Data is collected from medical record.
Incidence of transfer to higher-level care | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Any indication. Data is collected from medical record.
Incidence of major morbidity before discharge | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Composite outcome defined as any of the following morbidities: intraventricular haemorrhage grade III or IV, cystic periventricular leukomalacia, retinopathy of prematurity ≥ grade 3, or BPD at 36 weeks' postmenstrual age

OTHER OUTCOMES:
Adverse events | Before discharge (about 6-15 weeks)
  Suspected or confirmed adverse events. Reported by clinical investigators, staff or during video analysis.
Pain or discomfort, measured by a neonatal pain scale | During the procedure, an average of 5-10 minutes
  Prespecified video analysis for subsample of 50 patients per treatment arm
Duration of procedure | During the procedure, an average of 5-10 minutes
  Numerical variable (seconds). Prespecified video analysis for subsample of 50 patients per treatment arm
Duration of desaturation of SpO2 <80%, <60% and <40% during procedure | During the procedure, an average of 5-10 minutes
  Numerical variable (seconds). Prespecified video analysis for subsample of 50 patients per treatment arm
Duration of heart rate <100 bpm and <60 bpm during procedure | During the procedure, an average of 5-10 minutes
  Numerical variable (seconds). Prespecified video analysis for subsample of 50 patients per treatment arm
Adherence to intervention protocol | During the procedure, an average of 5-10 minutes
  Categorical variable (Yes/No). Adherence to intervention proctol for SALSA or INSURE. Prespecified video analysis for subsample of 50 patients per treatment arm.
Pilot outcome: Recruitment rate | At randomization.
  Numerical variable. Number of patients enrolled in the trial per month.
Pilot outcome: Adherence to assigned intervention | After procedure, approximately 5-10 minutes
  Categorical variable (Yes/No). Infant receiving the assigned surfactant method.
  - Comparing proportion between arms.
Pilot Outcome: Adherence to invasive mechanical ventilation criteria | Until 72 hours after first surfactant administration
  Categorical variable (Yes/No). Did infant have a documented clinical indication for mechanical ventilation, as per local NICU criteria, if received invasive mechanical ventilation within 72 hours of randomization.
  * Comparing proportion between arms.
  * Differences in indication for mechanical ventilation between study arms will be explored descriptively.
Pilot Outcome: Attrition rate | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Defined as withdrawal from the study or loss to follow-up before outcomes can be assessed
Pilot Outcome: Data completeness | Before discharge (about 6-15 weeks)
  Categorical variable (Yes/No). Missing primary or secondary outcomes. Comparing proportion between arms.
Pilot Outcome: Data integrity | Before discharge (about 6-15 weeks)
  Numerical variable. Defined as the consistency between recorded trial data and source data, as determined through source data verification according to the monitoring plan. Measured as number of inconsistent data fields. Proportion of inconsistent fields to be compared between arms.
Pilot Outcome: Acceptability of SALSA | Before discharge (about 6-15 weeks)
  Based on a survey to staff and parents, in beginning and end of pilot phase

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Alfvén, Professor, M.D, Ph.D, Principal Investigator — Department of Global Public Health, Karolinska Institutet, Solna, Sweden
Locations (1):
- Phu San Hanoi Hospital - Hanoi Obstetrics and Gynecology Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request after publication of results.
Supporting Information: Study Protocol, ICF
Time Frame: Can be available from the principal investigator on reasonable request
Access Criteria: Can be available from the principal investigator on reasonable request

REFERENCES:
- [Background] Zapata HA, Fort P, Roberts KD, Kaluarachchi DC, Guthrie SO. Surfactant Administration Through Laryngeal or Supraglottic Airways (SALSA): A Viable Method for Low-Income and Middle-Income Countries. Front Pediatr. 2022 Mar 16;10:853831. doi: 10.3389/fped.2022.853831. eCollection 2022. PMID 35372140
- [Background] Dempsey T, Brismar TB, Svensson-Marcial A, Blennow M, Alfven T, Hook SM, Pejovic N. Radiologic evaluation of three smaller-sized supraglottic airway device prototypes for low-birth-weight neonates. Br J Anaesth. 2025 Nov;135(5):1551-1553. doi: 10.1016/j.bja.2025.05.038. Epub 2025 Jul 3. No abstract available. PMID 40610284
- [Background] Abdel-Latif ME, Walker E, Osborn DA. Laryngeal mask airway surfactant administration for prevention of morbidity and mortality in preterm infants with or at risk of respiratory distress syndrome. Cochrane Database Syst Rev. 2024 Jan 25;1(1):CD008309. doi: 10.1002/14651858.CD008309.pub3. PMID 38270182
- See also: Feasibility study of SALSA using the same device at the same hospital in infants with birth weigh 750-1500g — https://www.clinicaltrials.gov/study/NCT06606444?cond=NCT06606444&rank=1